CLINICAL TRIAL: NCT05970861
Title: Effect of Natural Food on Gut Microbiome and Phospholipid Spectrum of Immune Cells in COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asfendiyarov Kazakh National Medical University (Other)
Responsible Party: Principal Investigator, Vildan Indershiyev, Ph.D. candidate, Asfendiyarov Kazakh National Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KazNMU_Saumal_COVID
Record Dates: First submitted 2023-07-31; First posted 2023-08-01 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: COVID-19
Keywords: COVID-19; gut microbiome; antiphospholipid antibodies; rehabilitation; food products
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Main Group (Experimental): Patients who had suffered from COVID-19 in the six months before the start of the study. Patients will receive Saumal (freeze-dried mare milk) for four weeks.
  Interventions: Dietary Supplement: Freeze-dried Mare Milk (Saumal)
- Control Group (No Intervention): Patients who had suffered from COVID-19 in the six months before the start of the study. There will be no intervention.

INTERVENTIONS:
Dietary Supplement: Freeze-dried Mare Milk (Saumal) — Freeze-dried Mare Milk (Saumal) is frequently reported for having therapeutic and dietary properties associated with specific chemical composition and certain physical properties of the product. It contains a total of about 40 biologically active components, the most important of them vitamins A, C, B1, B2, B6, and B12, amino acids, enzymes, and trace elements (low molecular weight peptides, lactalbumins, and globulins). Saumal will be administered to patients at a dose of 25 grams of dry powder per 200 ml of water, 2 times a day, 30 minutes before the meal, for 4 weeks.
  Arms: Main Group

SUMMARY:
The efficacy of natural foods such as freeze-dried mare's milk (Saumal) in post-COVID syndrome therapy has not been studied. The literature review has shown that researchers have focused more on evidence-based medications and less on natural products. Some raw foods, such as freeze-dried mare's milk, contribute to forming complete immune complexes and have antioxidant, membrane stabilizing, and antiviral effects.

The use of Saumal proved its effectiveness in patients suffering from chronic hepatitis C. After 4 weeks of using freeze-dried mare's milk, the biodiversity of the intestinal microbiome was increased. The content of bacteria secreting short-chain fatty acids also increased.

The study aims to confirm these effects at the gene level in patients who underwent COVID-19. This study will allow us to develop a highly evidence-based component of rehabilitation therapy in patients after COVID-19.

DETAILED DESCRIPTION:
The study consists of three stages. Stage I. Randomized division of 75 patients under study into a main group of 38 patients receiving Saumal for 4 weeks and a control group of 37 patients not receiving Saumal. All respondents have suffered from COVID-19 in the last 6 months. At the moment of the research, all patients will be staying in rehabilitation centers in Almaty City.

The study's biological material will be collected from the respondents (gut microbiome, antiphospholipid antibodies, biochemical blood analysis (glucose, ALT, AST, uric acid, TAGs, alkaline phosphatase)).

Stage II. The main group will be given Saumal for four weeks, after which the gut microbiome, antiphospholipid antibodies, and biochemical blood analysis will be collected from both groups again. This will allow us to assess the impact of freeze-dried mare's milk on the condition of the gut microbiome, antiphospholipid antibodies, and biochemical blood analysis.

Stage III. Data analysis.

1. Based on the results of gut microbiome sequencing, ELISA (antiphospholipid antibodies), and biochemical blood analysis in the main and control groups, we determine the dynamic changes of those parameters during COVID-19 rehabilitation.
2. According to the results, the effectiveness of Saumal itself regarding these 2 parameters will be evaluated.
3. Develop recommendations and an algorithm for patient management after COVID-19 to prevent complications.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older;
2. Patients in rehabilitation after COVID-19;
3. Signed informed consent;
4. Presence of patient's history of COVID-19, reliably established by PCR+ /presence of IgG/ diagnosis of coronavirus pneumonia on Computer Tomography based on discharge from hospital or outpatient records.

Exclusion Criteria:

1. Chronic inflammatory bowel disease;
2. Gut microbiota transplantation;
3. Chronic pancreatic disease, period of exacerbation;
4. Liver cirrhosis, Metavir stage 3-4;
5. Any disease in the decompensation stage;
6. Neuralgic and psychological disorders that interfere with the study;
7. Cancer;
8. Non-transportable patients;
9. Patients who do not reside in Almaty;
10. Patients who have refused to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ainur Yeshmanova, Ph.D., Study Director — Asfendiyarov Kazakh National Medical University; Nikolay Safonov, Study Chair — Asfendiyarov Kazakh National Medical University; Zhannat Nurmakhanova, Ph.D, Study Chair — Asfendiyarov Kazakh National Medical University; Zhanar Nurgaliyeva, Ph.D., Study Chair — Asfendiyarov Kazakh National Medical University
Locations (1):
- Almaty House of Veterans, Almaty, Kazakhstan

REFERENCES:
- [Background] Zuo T, Zhang F, Lui GCY, Yeoh YK, Li AYL, Zhan H, Wan Y, Chung ACK, Cheung CP, Chen N, Lai CKC, Chen Z, Tso EYK, Fung KSC, Chan V, Ling L, Joynt G, Hui DSC, Chan FKL, Chan PKS, Ng SC. Alterations in Gut Microbiota of Patients With COVID-19 During Time of Hospitalization. Gastroenterology. 2020 Sep;159(3):944-955.e8. doi: 10.1053/j.gastro.2020.05.048. Epub 2020 May 20. PMID 32442562
- [Background] Yeoh YK, Zuo T, Lui GC, Zhang F, Liu Q, Li AY, Chung AC, Cheung CP, Tso EY, Fung KS, Chan V, Ling L, Joynt G, Hui DS, Chow KM, Ng SSS, Li TC, Ng RW, Yip TC, Wong GL, Chan FK, Wong CK, Chan PK, Ng SC. Gut microbiota composition reflects disease severity and dysfunctional immune responses in patients with COVID-19. Gut. 2021 Apr;70(4):698-706. doi: 10.1136/gutjnl-2020-323020. Epub 2021 Jan 11. PMID 33431578
- [Background] Romaniuk K., Majszyk-Świątek M., Kryszak K., Danielewicz A., Andraszek K. Alternative use of mare milk. Folia Pomer. Univ. Technol. Stetin. 2019;348:121-130. doi: 10.21005/AAPZ2019.49.1.13.
- [Background] Kushugulova A., Kozhakhmetov S., Sattybayeva R., Nurgozhina A., Ziyat A., Yadav H., Marotta F. Mare's milk as a prospective functional product. Funct. Food Health Dis. 2018;8:537-543. doi: 10.31989/ffhd.v8i11.528.
- [Background] Musayev, A., Yeshmanova, A., Pakhomenko, Y., Kozhakhmetov, S.S., Kushugulova, A.K. Effects of Environmental Pollutants on Intestinal Microbiome Under the Influence Of Mare's Milk In Patients with Hepatitis C. Procedia Environmental Science, Engineering and Management 2020;7(4):605-611.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Main Group | Control Group
Started | 38 (Originally, we planned to include 38 patients in the main group and 37 in the control group. Overall, these groups were evenly divided, with 30 patients in each group.) | 37 (Originally, we planned to include 38 patients in the main group and 37 in the control group. Overall, these groups were evenly divided, with 30 patients in each group.)
Completed | 30 (Originally, we planned to include 38 patients in the main group and 37 in the control group. Overall, these groups were evenly divided, with 30 patients in each group.) | 30 (Originally, we planned to include 38 patients in the main group and 37 in the control group. Overall, these groups were evenly divided, with 30 patients in each group.)
Not Completed | 8 | 7
Not completed — Physician Decision | 4 | 4
Not completed — Lost to Follow-up | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Group | Control Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 10 | 10 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 10 | 10 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Count of Participants [Count of Participants; unit: Participants] | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Gut Microbiome
Description: Intestinal microbiome studies will be performed using the Illumina MiSeq Metagenomics Kit. Creation of libraries for NGS sequencing. The commercial Illumina MiSeq The Metagenomics Kit includes two primer pools that can amplify the hypervariable regions of 16S rRNA in bacteria. The first pool produces V2-4-8, while the second pool allows for the production of V3-6 and 7-9 regions of 16S rRNA. Sequencing will be performed on an Ion S5 analyzer using an Illumina MiSeq Chip Kit. Once the PCR products have been run, it is important to follow standard procedures for fragment end recovery, adaptor ligation, nick gap repair, qualitative and quantitative assessment of non-amplified libraries, and pooling.
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: Mean percentages of gut microbiota units
Arm/Group | Main Group | Control Group
Number analyzed (Participants) | 30 | 30
Mean percentages of gut microbiota units
  Percentage of "Firmicutes" phylum at 4 weeks | 51.87 (0.001) | 46.1 (0.899)
  Percentage of "Bacteroides" phylum at 4 weeks | 29.43 (0.178) | 29.77 (0.754)
  Percentage of "Proteobacteria" phylum at 4 weeks | 6.52 (0.00001) | 7.91 (0.823)
  Percentage of "Actinobacteria" phylum at 4 weeks | 4.9 (0.951) | 9.36 (0.003)
  Percentage of "Bacilli" class at 4 weeks | 4.02 (0.043) | 4.46 (0.068)
  Percentage of "Deltaproteobacteria" class at 4 weeks | 0.94 (0.048) | 0.92 (0.918)
  Percentage of "Erysipelotrichi" class at 4 weeks | 1.58 (0.012) | 1.46 (0.889)
  Percentage of "Caldilinea" genus at 4 weeks | 0.06 (0.014) | 0.17 (0.345)
  Percentage of "Clostridium" genus at 4 weeks | 5.07 (0.008) | 2.59 (0.893)
  Percentage of "Desulfovibrio" genus at 4 weeks | 0.19 (0.039) | 0.76 (0.008)
  Percentage of "Escherichia" genus at 4 weeks | 0.75 (0.042) | 1.2 (0.710)
  Percentage of "Lachnospira" genus at 4 weeks | 1.77 (0.004) | 1.76 (0.049)
  Percentage of "Prevotella" genus at 4 weeks | 8.85 (0.003) | 11.24 (0.698)
  Percentage of "Tindallia" genus at 4 weeks | 0.20 (0.02) | 0.00 (1.00)
  Percentage of "Anaerobranca zavarzinii" species at 4 weeks | 0.62 (0.006) | 0.18 (0.004)
  Percentage of "Alkaliphilus crotonatoxidans" species at 4 weeks | 1.40 (0.00001) | 0.93 (0.028)
  Percentage of "Bacteroides xylanisolvens" species at 4 weeks | 1.30 (0.00001) | 1.63 (0.245)
  Percentage of "Bifidobacterium catenulatum" species at 4 weeks | 0.96 (0.024) | 1.68 (0.434)
  Percentage of "Bifidobacterium indicum" species at 4 weeks | 0.10 (0.026) | 0.20 (0.052)
  Percentage of "Roseburia faecis" species at 4 weeks | 0.72 (0.006) | 0.36 (0.551)
Statistical Analysis 1: Comparison: Main Group vs Control Group; Null hypothesis: there is no statistical significance between the mean percentages of microbiota units of the main and control groups after the mare's milk administration. Alternate hypothesis: statistical significance exists between the mean percentages of microbiota units of the main and control groups after the mare's milk administration; Test type: Other; p < 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Main Group vs Control Group; Null Hypothesis: The freeze-dried mare's milk does not significantly influence the mean percentages of gut microbiota units. Alternate Hypothesis: The freeze-dried mare's milk significantly influences the mean percentages of gut microbiota units; Test type: Other; p < 0.05, ANOVA

2. Primary Outcome: Antiphospholipid Antibodies
Description: IgG or IgM autoantibodies to cardiolipin, phosphatidyl serine, phosphatidyl-inositol, phosphatidyl acid, and β2-glycoprotein I are determined in human venous blood serum by enzyme immunoassay (ELISA) using the Anti-Phospholipid Screen IgG/IgM kit.
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: U/ml
Arm/Group | Main Group | Control Group
Number analyzed (Participants) | 30 | 30
U/ml
  IgM | 2.73 (0.185) | 4.45 (0.001)
  IgG | 1.43 (0.726) | 4.50 (0.0001)
Statistical Analysis 1: Comparison: Main Group vs Control Group; Null hypothesis: No statistically significant difference exists between antiphospholipid antibody levels before and after the mare's milk administration. Alternate hypothesis: Statistically significant difference exists between antiphospholipid antibody levels before and after the mare's milk administration; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Biochemical Blood Analysis (Uric Acid)
Description: This biochemical indicator will be determined from patient serum on a BA400 analyzer (BioSystems S.A., Spain)
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Main Group | Control Group
Number analyzed (Participants) | 30 | 30
mg/dL | 5.56 (0.01) | 7.87 (0.34)
Statistical Analysis 1: Comparison: Main Group vs Control Group; Null hypothesis: No statistically significant difference exists between uric acid blood levels before and after the mare's milk administration. Alternate hypothesis: Statistically significant difference exists between uric acid blood levels before and after the mare's milk administration; Test type: Other; p = 0.01, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Quality of Life Changes
Description: Constructs: Physical Functioning (PF), Role Limitations due to Physical Health (RP), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Functioning (SF), Role Limitations due to Emotional Problems (RE), Mental Health (MH). All scale ranges (for any construct): 0 to 100.
  Higher scores indicate: PF - better physical functioning; RP - fewer role limitations due to physical health; BP - less bodily pain; GH - better perceived general health; VT - greater vitality and less fatigue; SF - better social functioning; RE - fewer role limitations due to emotional problems; MH - better mental health.
  The SF-36 does not have a single total score but can be summarized using two summary measures:
  1. Physical Component Summary (PCS). Combines the following scales: PF, RP, BP, GH.
  2. Mental Component Summary (MCS). Combines the following scales: VT, SF, RE, MH. Higher scores indicate better physical and mental health. Range: Typically standardized (mean = 50, SD = 10)
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Main Group | Control Group
Number analyzed (Participants) | 30 | 30
T-score
  PCS | 47.965 (0.004) | 50.797 (0.647)
  MCS | 49.524 (0.001) | 49.393 (0.091)
Statistical Analysis 1: Comparison: Main Group; Null hypothesis: No statistically significant difference exists between the scores on a scale (PCS, MCS) after the mare's milk administration. Alternate hypothesis: Statistically significant difference exists between the scores on a scale (PCS, MCS) after the mare's milk administration; Test type: Other; p < 0.01, t-test, 2 sided
Statistical Analysis 2: Comparison: Control Group; Null hypothesis: No statistically significant difference exists between the scores on a scale (PCS, MCS) after 2 measurements in the control group. Alternate hypothesis: Statistically significant difference exists between the scores on a scale (PCS, MCS) after 2 measurements in the control group; Test type: Other; p > 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: Main Group vs Control Group; Null Hypothesis: The freeze-dried mare's milk does not significantly influence the scores on the scales (PCS, MCS). Alternate Hypothesis: The freeze-dried mare's milk significantly influences the scores on the scales (PCS, MCS); Test type: Other; p < 0.01, ANOVA

5. Secondary Outcome: Biochemical Blood Analysis (ALT)
Description: This biochemical indicator will be determined from patient serum on a BA400 analyzer (BioSystems S.A., Spain)
Time Frame: 4 weeks
Measure: Mean (Full Range); unit: units per liter (IU/L)
Arm/Group | Main Group | Control Group
Number analyzed (Participants) | 30 | 30
units per liter (IU/L) | 31 [25 to 37] | 35 [23 to 47]

6. Secondary Outcome: Biochemical Blood Analysis (AST)
Description: This biochemical indicator will be determined from patient serum on a BA400 analyzer (BioSystems S.A., Spain)
Time Frame: 4 weeks
Measure: Mean (Full Range); unit: units per liter (IU/L)
Arm/Group | Main Group | Control Group
Number analyzed (Participants) | 30 | 30
units per liter (IU/L) | 34 [25 to 43] | 33 [27 to 39]

7. Secondary Outcome: Biochemical Blood Analysis (Glucose)
Description: This biochemical indicator will be determined from patient serum on a BA400 analyzer (BioSystems S.A., Spain)
Time Frame: 4 weeks
Measure: Mean (Full Range); unit: mmol/L
Arm/Group | Main Group | Control Group
Number analyzed (Participants) | 30 | 30
mmol/L | 5.4 [4.2 to 6.6] | 5.7 [3.8 to 7.6]

8. Secondary Outcome: Biochemical Blood Analysis (Triacylglycerides)
Description: This biochemical indicator will be determined from patient serum on a BA400 analyzer (BioSystems S.A., Spain)
Time Frame: 4 weeks
Measure: Mean (Full Range); unit: mmol/L
Arm/Group | Main Group | Control Group
Number analyzed (Participants) | 30 | 30
mmol/L | 1.5 [1.3 to 1.7] | 1.4 [1.2 to 1.6]

9. Secondary Outcome: Biochemical Blood Analysis (Alkaline Phosphatase)
Description: This biochemical indicator will be determined from patient serum on a BA400 analyzer (BioSystems S.A., Spain)
Time Frame: 4 weeks
Measure: Mean (Full Range); unit: IU/L
Arm/Group | Main Group | Control Group
Number analyzed (Participants) | 30 | 30
IU/L | 85 [65 to 105] | 92 [70 to 114]

ADVERSE EVENTS:
Time Frame: Any adverse events have not been monitored or evaluated.
Description: Any adverse events have not been monitored or evaluated.
Arm/Group | Main Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
There were three main limitations to the study:

1. A significant amount of time has passed since the patients had COVID-19.
2. During the analysis of antiphospholipid antibody levels, we found that screening kits were used.
3. The severity of COVID-19 was not considered as an inclusion criterion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT05970861/Prot_SAP_000.pdf